CLINICAL TRIAL: NCT01986803
Title: Comparison of the ABSORBTM Everolimus Eluting Bioresorbable Vascular Scaffold System With a Drug- Eluting Metal Stent (XienceTM) in Acute ST-Elevation Myocardial Infarction
Brief Title: ABSORB STEMI: the TROFI II Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Abbott Medical Devices (Industry); Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECRI-003
Record Dates: First submitted 2013-08-29; First posted 2013-11-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
Keywords: ST-elevation Myocardial Infarction (STEMI); Primary Percutaneous Coronary Intervention within 24 hrs; Healing score; OFDI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI with ABSORBTM bioresorbable vascular scaffold system (BVS) (Experimental): All patients assigned to the experimental arm will be treated with a primary Percutaneous Coronary Intervention using the Abbott Vascular ABSORB TM everolimus eluting bioresorbable vascular scaffold system (BVS)
  Interventions: Device: Percutaneous Coronary Intervention
- PCI with XIENCE Xpedition stent (Active Comparator): All patients assigned to the experimental arm will be treated with a primary Percutaneous Coronary Intervention using the XIENCE Everolimus Eluting Coronary Stent System (XIENCE Xpedition) (commercial product)
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Implanting a device ("Xience Xpedition" stent or "Abbott Vascular ABSORBTM everolimus eluting bioresorbable vascular scaffold system (BVS)" to open a diseased coronary artery by going to the coronary artery subcutaneously through the arteries from the radial or femoral artery access point.

SUMMARY:
This is a Prospective, randomized (1:1), active control, single-blind, non-inferiority, European multicenter clinical trial.

The primary objective of this study is to assess the neointimal healing score (as evaluated by intra-coronary OFDI) in patients with ST-elevation Myocardial Infarction (STEMI) and treated with Abbott Vascular ABSORB everolimus eluting bioresorbable vascular scaffold (BVS) at 6 months follow-up by comparing with a metallic drug eluting stent (XIENCE). Furthermore, the safety and feasibility of implanting ABSORB BVS in patients with STEMI is assessed.

It is hypothesized that acutely and at 6 months follow-up implantation of the ABSORB fully bioresorbable everolimus-eluting scaffold is at least as safe as implantation of metallic drug-eluting stent, and that at late follow-up the ABSORB scaffold could improve the arterial healing process and potentially reduce late stent thrombosis in patients presenting with STEMI.

This is a preparatory trial in anticipation of a major outcome study.

DETAILED DESCRIPTION:
A total of 190 patients will be included in this trial, at 8-10 European sites.

The primary endpoint is arterial healing at 6 month follow up. To assess the arterial healing, at 6 months follow-up all patients will undergo angiographic follow-up with OFDI investigation. To score the arterial healing, a Healing Score is used.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age;
2. Primary PCI within 24 hours of symptom onset;
3. ST-segment elevation of > 1mm in > 2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of >1mm in >2 contiguous anterior leads;
4. Presence of at least one acute infarct artery target vessel with one or more coronary artery stenoses in a native coronary artery within planned device deployment segment (Dmax) by visual estimation of ≥ 2.5 mm and ≤ 3.8 mm;
5. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 6 months following the index procedure.

Exclusion Criteria:

1. Inability to provide informed consent;
2. Known pregnancy at time of randomization. Female who is breastfeeding at time of randomization;
3. Known intolerance to aspirin, heparin, PLLA (poly(L-lactic acid), everolimus, contrast material;
4. Cardiogenic Shock;
5. Unprotected left main coronary artery stenosis;
6. Distal occlusion of target vessel;
7. Acute myocardial infarction secondary to stent thrombosis;
8. Mechanical complications of acute myocardial infarction;
9. Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in sub-optimal imaging or excessive risk of complication from placement of an OFDI catheter;
10. Fibrinolysis prior to PCI;
11. Active bleeding or coagulopathy or patients at chronic anticoagulation therapy;
12. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Healing Score | 6 months follow-up
  The primary endpoint is: Healing Score at 6 months follow-up. This is measured with OFDI imaging.
  This Healing Score is a weighted index that combines the following parameters:
  1. Presence of filling defect (%ILD) is assigned weight of "4",
  2. Presence of both malapposed and uncovered struts (%MN) is assigned a weight of "3",
  3. Presence of uncovered struts alone (%N) is assigned a weight of "2" and finally,
  4. Presence of malapposition alone (%M) is assigned a weight of "1".

SECONDARY OUTCOMES:
Procedure success | Study patients will be followed for the duration of hospital stay (e.g. until hospital discharge), an expected average of 2 days.
  Clinical Endpoint. Procedure success is no in-hospital Device Oriented Composite Endpoint, which is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Device-Oriented Composite Endpoint | Up to 3 years
  Clinical Endpoint. Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Cardiac Death | Up to 6 months
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
Cardiac Death | Up to 3 years
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
MI not clearly attributable to a non-intervention vessel | Up to 6 months
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
MI not clearly attributable to a non-intervention vessel | Up to 3 years
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
Clinically-indicated target lesion revascularization | Up to 6 months
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
Clinically-indicated target lesion revascularization | Up to 3 years
  Clinical Endpoint. One of the individual components of the Device Oriented Composite Endpoints, which is a secondary endpoint on itself.
All-cause death at all timepoints | Up to 6 months
  Clinical Endpoint.
All-cause death at all timepoints | Up to 3 years
  Clinical Endpoint.
Any Myocardial Infarction at all timepoints | Up to 6 months
  Clinical Endpoint.
Any Myocardial Infarction at all timepoints | Up to 3 years
  Clinical Endpoint.
Non Ischemia-driven target lesion revascularization (TLR) at all timepoints | Up to 6 months
  Clinical Endpoint.
Non Ischemia-driven target lesion revascularization (TLR) at all timepoints | Up to 3 years
  Clinical Endpoint.
Ischemia-driven and non ischemia-driven target vessel revascularization (TVR) at all timepoints | Up to 6 months
  Clinical Endpoint.
Ischemia-driven and non ischemia-driven target vessel revascularization (TVR) at all timepoints | Up to 3 years
  Clinical Endpoint.
Scaffold/Stent thrombosis according to ARC definitions at all timepoints | Up to 6 months
  Clinical Endpoint. ARC = academic research consortium
Scaffold/Stent thrombosis according to ARC definitions at all timepoints | Up to 3 years
  Clinical Endpoint. ARC = academic research consortium
Angina Class at all timepoints | Up to 6 months
  Clinical Endpoint. Angina Pectoris
Angina Class at all timepoints | Up to 3 years
  Clinical Endpoint. Angina Pectoris
Other Serious Adverse Events at all timepoints | Up to 6 months
  Clinical Endpoint.
Other Serious Adverse Events at all timepoints | Up to 3 years
  Clinical Endpoint.
Device-Oriented Composite Endpoint | Up to 6 months
  Clinical Endpoint. Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Percent diameter stenosis (%DS) | Up to 6-months
  Angiographic endpoint. Percent diameter stenosis (%DS)at in in-segment (target lesion), in-device, proximal and distal
Minimal Lumen Diameter(MLD) | Up to 6-months
  Angiographic endpoint. Minimal Lumen Diameter(MLD)at in in-segment (target lesion), in-device, proximal and distal
Late loss of the target lesion | Up to 6-months
  Angiographic endpoint. Late loss (LL), which is decrease in blood vessel lumen diameter, at in in-segment (target lesion), in-device, proximal and distal
Angiographic binary restenosis (ABR) | Up to 6-months
  Angiographic endpoint. Angiographic binary restenosis (ABR)at in in-segment (target lesion), in-device, proximal and distal
Presence of filling defect (%ILD) | 6-months
  OFDI endpoint. Presence of filling defect (%ILD), which is an individual component of the primary endpoint "Healing Score".
Presence of both malapposed and uncovered struts (%MN) | 6-months
  OFDI endpoint. Presence of both malapposed and uncovered struts (%MN)of the index stent, which is an individual component of the primary endpoint "Healing Score".
Presence of uncovered struts alone(%N) | 6-months
  OFDI endpoint. Presence of both uncovered struts of the index stent, which is an individual component of the primary endpoint "Healing Score".
Presence of malapposed struts alone(%M) | 6-months
  OFDI endpoint. Presence of both malapposed struts of the index stent, which is an individual component of the primary endpoint "Healing Score".
Mean/minimal scaffold/stent diameter/area/volume | 6-months
  OFDI endpoint. Mean/minimal scaffold/stent diameter/area/volume at 6-months follow-up.
Mean/minimal lumen diameter/area/volume | 6-months
  OFDI endpoint. Mean/minimal lumen diameter/area/volume at 6-months follow-up.
Incomplete strut apposition (ISA) area/volume | 6-months
  OFDI endpoint. Incomplete strut apposition (ISA) area/volume at 6-months follow-up.
Percentage of covered struts | 6-months
  OFDI endpoint. Percentage of covered struts at 6-months follow-up.
Mean/maximal thickness of the struts coverage | 6-months
  OFDI endpoint. Mean/maximal thickness of the struts coverage at 6-months follow-up.
Neointimal hyperplasia area/volume | 6-months
  OFDI endpoint. Neointimal hyperplasia area/volume at 6-months follow-up.
Mean Flow area/volume | 6-months
  OFDI endpoint. Mean Flow area/volume at 6-months follow-up.
Intraluminal defect area/volume | 6-months
  OFDI endpoint. Intraluminal defect area/volume at 6-months follow-up.
Thickness of neointimal tissue developed over lipid rich plaque | 6-months
  OFDI endpoint. Thickness of neointimal tissue developed over lipid rich plaque at 6-months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: P. Serruys, Prof., Principal Investigator — Erasmus Medical Centre Rotterdam, the Netherlands; M. Sabaté, Dr., Principal Investigator — University of Barcelona, Spain; S. Windecker, Dr., Principal Investigator — Bern University Hospital, Bern, Switzerland
Locations (8):
- Denmark (2):
  - Research centre Aarhus, DK003, Aarhus
  - Research centre Odense, DK002, Odense
- Netherlands (2):
  - Research centre Leeuwarden, NL002, Leeuwarden
  - Research centre Nieuwegein, NL014, Nieuwegein
- Spain (3):
  - Research centre Barcelona, ES001, Barcelona
  - Research centre Barcelona, ES003, Barcelona
  - Research centre Vigo, ES004, Vigo
- Research centre Bern, CH006, Bern, Switzerland

REFERENCES:
- [Derived] Cassese S, Katagiri Y, Byrne RA, Brugaletta S, Alfonso F, Raber L, Maeng M, Iniguez A, Kretov E, Onuma Y, Joner M, Sabate M, Laugwitz KL, Windecker S, Kastrati A, Serruys PW. Angiographic and clinical outcomes of STEMI patients treated with bioresorbable or metallic everolimus-eluting stents: a pooled analysis of individual patient data. EuroIntervention. 2020 Mar 20;15(16):1451-1457. doi: 10.4244/EIJ-D-18-01080. PMID 30719976
- [Derived] Yamaji K, Brugaletta S, Sabate M, Iniguez A, Jensen LO, Cequier A, Hofma SH, Christiansen EH, Suttorp M, van Es GA, Sotomi Y, Onuma Y, Serruys PW, Windecker S, Raber L. Effect of Post-Dilatation Following Primary PCI With Everolimus-Eluting Bioresorbable Scaffold Versus Everolimus-Eluting Metallic Stent Implantation: An Angiographic and Optical Coherence Tomography TROFI II Substudy. JACC Cardiovasc Interv. 2017 Sep 25;10(18):1867-1877. doi: 10.1016/j.jcin.2017.07.035. PMID 28935079
- See also: Primary endpoint manuscript (PUBMED ID: 26405232) — https://www.ncbi.nlm.nih.gov/pubmed/26405232